CLINICAL TRIAL: NCT07020260
Title: The PACMAN-hu19 Trial: a Phase I/II Study to Investigate the Safety and Feasibility of Point-of-care Human CD19 Targeting CAR T-cells in Pediatric and Young Adult Patients With Relapsed or Refractory B-cell Malignancies
Brief Title: The PACMAN-Hu19 Trial: a Study of the Safety and Feasibility of Locally Produced, CD19-targeted and Human CAR T-cell Therapy in Children and Young Adults With Relapsed or Refractory B-cell Malignancies
Acronym: PACMAN
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Princess Maxima Center for Pediatric Oncology (Other)
Collaborators: Dutch Cancer Society (Other); Miltenyi Biomedicine GmbH (Industry); University Medical Center Utrecht (UMCU) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2023-507597-40; 2023-507597-40-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-26; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Leukemia; Lymphoma
Keywords: CAR T-cell Therapy; relapsed B-cell malignancies; refactory B-cell malignancies; B-NHL; B-cell ALL
MeSH Terms: conditions — Leukemia; Lymphoma; Burkitt Lymphoma | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Intervention Model Description: Each subject will receive a single infusion of the huCAR19 CAR T-cells. There will be 3 different dose levels investigated in the PACMAN trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- huCAR19 T-cells (Experimental): Participants will receive one single dose of huCAR19 T-cell infusion on day 0 of the treatment.
  Interventions: Other: CAR T-cell and Cellular Therapies

INTERVENTIONS:
Other: CAR T-cell and Cellular Therapies — A single IV infusion of huCAR 19 T-cells on day 0. In phase I 3 dose levels are tested to determine the RP2D.

SUMMARY:
PACMAN is a phase I/II single arm, open-label, multi-center study evaluating the safety of human CD19 CAR-T (huCAR19) produced locally using the Miltenyi Prodigy in children, adolescents and young adults with relapsed/refractory CD19+ hematological malignancies for whom no standard of care treatment is available.

DETAILED DESCRIPTION:
In this study patients aged 1-45 years with relapsed or refractory CD19+ hematological malignancies (B-NHL or BCP-ALL) are treated with a single dose of huCAR19 T-cells. After consent and screening, patients will undergo leukapheresis to harvest autologous PBMCs. During the CAR T-cell production, patients receive lymphodepleting chemotherapy after which the huCAR19 T-cells are administered. In phase I the aim is to establish the RP2D, the protocol will then be extended to a phase II.

ELIGIBILITY:
Inclusion Criteria:

1. 1-45 years of age.
2. Patients with relapsed or refractory CD19+ hematological malignancies including, but not limited to:

   1. B-NHL such as Burkitt lymphoma(BL), de novo or transformed diffuse large B cell lymphoma (DLBCL), lymphoblastic lymphoma (LBL), primary mediastinal B cell lymphoma (PMBCL) or indolent lymphoma types with no access to commercially available CAR T-cell therapy or for whom the current production time for commercially available CAR T-cell therapy is not acceptable based on medical need.

      OR
   2. B-cell precursor ALL failing commercially available CAR T-cell therapy, or for BCP-ALL indications with no access to commercially available CAR T-cell therapy, or for whom the current production time for commercially available CAR T-cell therapy is not acceptable based on urgent medical need (the latter needs to be confirmed by the sponsor).
3. Measurable disease:

   1. For B-NHL at least one measurable lesion according to the Lugano classification.
   2. For BCP-ALL at least 0.1% (=10-3) of blasts should be present in the bone marrow measured by molecular MRD, morphology or flow cytometry at screening.
4. Patients must have exhausted or are ineligible for all registered therapeutic options with curative potential.
5. Adequate performance score:

   1. Children <16 years: Lansky performance status ≥ 60 .
   2. Children age ≥16 years and <18 years Karnofsky performance status ≥ 60.
   3. Adults ≥18 years ECOG performance status 0, 1 or 2 (ECOG performance status 3 is allowed only when due to underlying disease).
6. Patients from childbearing potential must be willing and able to use highly effective methods of birth control from first chemotherapy infusion through 12 months after administering the last study treatment.
7. Patients must be willing to abstain from breast feeding through 12 months after administering the last study treatment.
8. Patients must agree to refrain from donating blood or organs following treatment with huCAR19 T-cells.
9. Written informed consent per local law and regulations.

   Additional inclusion criteria phase I part of the study:
10. The first three patients in the phase I part of the study must be aged 12-45 years, thereafter patients of any age between 1-45 years can be recruited once surrogate endpoint of BCA is reached in ≥60% patients in previous or current dose level and ≤1 DLT occurred at the previous dose level.

Exclusion Criteria:

1. Patients with symptomatic CNS involvement will be excluded. After resolution and control of symptoms, patients can be rescreened.
2. Active uncontrolled or life-threatening infections.
3. Infection with HTLV-1, HTLV-2, HIV-1, HIV-2, hepatitis B (HbsAg positive) or hepatitis C (anti-HCV positive). Chronic controlled hepatitis B or C infection with undetectable viral load or controlled HIV infection with viral load <50 IU/ml and CD4+ T-cell count >200/ml may be considered when antiviral prophylaxis or therapy can be administered.
4. Absolute neutrophil count <0.5x109/L unless caused by underlying disease.
5. Platelet count <25x109/L unless caused by underlying disease.
6. Bilirubin and/or transaminases ≤ 2.5 x ULN, unless caused by underlying disease.
7. Renal insufficiency, defined as:

   1. For adults (≥18 years) glomerular filtration rate (GFR) < 45 ml/min/1.73 m2 as calculated by the Modification of Diet in Renal Disease (MDRD) equation:

      predicted GFR (ml/min/1.73 m2) = 186 x (serum creatinine in umol/L / 88.7) - 1.154 x (age in years) - 0.203 x (0.742 if patient is female) x (1.212 if patient is black).
   2. For children (<18 years) a serum creatinine based on gender/age as follows (in µmol/l):

   Age Male Female 0 to < 2 years 53 70 2 to < 6 years 70 70 6 to < 10 years 88 88 10 to < 13 years 106 106 13 to < 16 years 132 123 16 to < 19 years 150 123
8. Inadequate pulmonary function defined as baseline oxygen saturation <92%, if not caused by underlying disease.
9. Inadequate cardiac function:

   1. Unstable angina or unstable cardiac arrhythmias.
   2. NYHA classification >II.
   3. LVSF <28% or LVEF <45% confirmed by echocardiogram or MUGA scan.
10. Concurrent malignancy requiring treatment of having been treated <3 months before screening except for curatively treated basal cell carcinoma of the skin.
11. Pregnant women.
12. Patients unable to participate in the study according to investigator judgement.
13. Patients not willing or unable to adhere to protocol guidelines or follow-up.
14. Treatment with allogeneic stem cell transplantation <12 weeks from screening or DLI <4 weeks from screening or active GVHD requiring systemic treatment. Cutaneous GVHD requiring only topical steroids is allowed.
15. Hypersensitivity to the active substance

Ages: 1 Year to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose (RP2D) | Within 28 days after huCAR19 infusion.
  The endpoint to measure this primary objective is the incidence of dose limiting toxicities (DLTs).

SECONDARY OUTCOMES:
To assess preliminary activity at day 28 for the BCP-ALL cohort and the overall response rate for the B-NHL cohort | For BCP-ALL: at day 28. For B-NHL: at day 90.
  For BCP-ALL: the MRD-negative CR rate. For B-NHL: the overall response rate (ORR, CR +PR according to Lugano criteria).
Duration of response, including the duration of B-cell aplasia | from inclusion through study completion
  Number of days until relapse. Number of days until loss of B-cell aplasia defined by ≥ 5 B-cells/µl.
Survival estimates. | Measured at 6 and 12 months.
  Event free survival (EFS); Overall survival (OS); Cumulative Incidence of Relapse (CIR).
The feasibility to produce HuCAR19 in the target population. | From day -13 (start of manufacturing) to day 0 (final analysis)
  Percentage of products fulfilling the release criteria.

OTHER OUTCOMES:
To assess protein levels during treatment including cytokines reported to correlate with specific adverse events of interest of CAR T-therapy, namely CRS and ICANS | during treatment
  Protein expression.
To assess anti-CAR T-immune responses. | From infusion to 12 months after infusion.
  Antibody formation and changes in immune cell subsets.
Extensive characterization of apheresis product, CAR T-product, and persisting CAR T-cells after infusion | From leukapheresis to 12 months after infusion.
  Immunophenotype of apheresis product, CAR T-product and persisting CAR T-cells after infusion.
  CAR T-cell expansion (peak expansion, AUC of first 28 days).
Measure levels of fludarabine during the lymphodepleting regimen | On day -5 and day -3 of treatment.
  Measure levels of fludarabine in peripheral blood.
Percentage of participating patients that experience improvement in their quality of life (QoL). | From screening to 12 months after infusion.
  Questionnaires are completed to determine improvement in QoL
Clinical burden: duration of hospitalization and re-admission | From informed consent to 12 months after infusion.
  Number of days in the hospital.
Financial burden | Day -21 until day 180.
  Costs of the production and treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Friso Calkoen, MD, PhD, Principal Investigator — Princess Maxima Center for Pediatric Oncology
Locations (2):
- Netherlands (2):
  - University Medical Center Utrecht, Utrecht, Utrecht
  - Princess Máxima Center for pediatric oncology, Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No
Only IPD used in the results publication.